CLINICAL TRIAL: NCT05987371
Title: Randomized, Double-blind, Placebo-controlled, Dose Exploration, Multicenter Phase II Clinical Trial to Evaluate the Efficacy and Safety of TQC3721 Suspension for Inhalation in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease.
Brief Title: A Clinical Trial of TQC3721 Suspension for Inhalation in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC3721-II-02
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TQC3721 Suspension for Inhalation (Twice a day)+ Salbutamol (Experimental): TQC3721 suspension for inhalation, twice a day for 4 weeks, Salbutamol sulfate inhalation aerosol is used as required.
  Interventions: Drug: TQC3721 suspension for inhalation; Drug: Salbutamol sulfate inhalation aerosol
- TQC3721 Suspension for Inhalation (Once a day)+ Salbutamol (Experimental): TQC3721 suspension for inhalation, once a day for 4 weeks, Salbutamol sulfate inhalation aerosol is used as required.
  Interventions: Drug: TQC3721 suspension for inhalation; Drug: Salbutamol sulfate inhalation aerosol
- TQC3721 matching placebo for inhalation (Twice a day)+ Salbutamol (Placebo Comparator): TQC3721 suspension placebo for inhalation, twice a day for 4 weeks, Salbutamol sulfate inhalation aerosol is used as required.
  Interventions: Drug: TQC3721 matching placebo for inhalation; Drug: Salbutamol sulfate inhalation aerosol
- TQC3721 matching placebo for inhalation (once a day)+ Salbutamol (Placebo Comparator): TQC3721 suspension placebo for inhalation, once a day for 4 weeks, Salbutamol sulfate inhalation aerosol is used as required.
  Interventions: Drug: TQC3721 matching placebo for inhalation; Drug: Salbutamol sulfate inhalation aerosol

INTERVENTIONS:
Drug: TQC3721 suspension for inhalation — TQC3721 suspension for inhalation is a dual inhibitor targeting PDE3/4.
  Arms: TQC3721 Suspension for Inhalation (Once a day)+ Salbutamol; TQC3721 Suspension for Inhalation (Twice a day)+ Salbutamol
Drug: TQC3721 matching placebo for inhalation — Placebo without active substance.
  Arms: TQC3721 matching placebo for inhalation (Twice a day)+ Salbutamol; TQC3721 matching placebo for inhalation (once a day)+ Salbutamol
Drug: Salbutamol sulfate inhalation aerosol — Salbutamol is short-acting β2 receptor agonists.

SUMMARY:
This is a phase II clinical trial to evaluate the efficacy and safety of TQC3721 Suspension for Inhalation in patients with moderate to severe Chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent form before the study and fully understand the content, process, and potential adverse reactions of the experiment;
* Capable of using the study nebulizer correctly and complying with all study restrictions and procedures;
* Aged between 30 and 75 years old (Including critical values), both men and women;
* Body mass index(BMI) within the range of 18-30 kg/m2 (Including critical values);
* The subject has no pregnancy plan and voluntarily adopts effective contraceptive measures for at least one month from screening until the last use of the study drug;
* Diagnosed as a COPD patient according to the Global initiative for chronic obstructive lung disease (GOLD) 2023 standard, and had symptoms that met COPD for at least 1 year before screening;
* Able to conduct acceptable and repeatable lung function measurements;
* Clinical stability of COPD within 4 weeks before screening visit (V1) and between V1 visit and V2 visit;
* Long acting Bronchiectasis or short acting Bronchiectasis were not regularly used at least 14 days before screening visit (V1);
* Long acting Bronchiectasis can be stopped during the study until the end of the study, and short acting Bronchiectasis can be stopped at least 6 hours before the pulmonary function test;
* Meet the restrictions on combination medication and expect to maintain the restrictions during treatment;
* Current smoking or smoking history ≥ 10 pack years (smoking at least 20 cigarettes per day for 10 consecutive years or smoking at least 10 cigarettes per day for 20 consecutive years, former cigarette smokers must stop smoking>6 months before visit 1).

Exclusion Criteria:

* A history of life-threatening COPD, including hospitalization in an intensive care unit and/or the need for intubation.
* Acute exacerbations of COPD requiring oral or parenteral steroid treatment within 3 months before screening (V1) or before randomization (V2).
* Received inhaled corticosteroids (ICS) treatment within 4 weeks prior to screening.
* Have a history of hospitalization for COPD at least once within 6 months prior to screening.
* Antibiotic treatment for upper and/or lower respiratory tract infection within 6 weeks before screening or before randomized visit (V2). Note: Patients with a history of upper/lower respiratory tract infection within 6 weeks cannot participate in the test, but can be re-screened 6 weeks after the infection is cured.
* COVID-19:

  1. Suspected or confirmed COVID-19 infection during screening (V1), confirmed by the laboratory or based on the medical judgment of the researcher; Subjects who are known to have contact with COVID-19 positive patients. Note: Subjects should remain Asymptomatic for 14 days or more after exposure, and only after being approved by the investigator can they be re-screened.
  2. Known COVID-19 infection history within 4 weeks before screening (V1);
  3. Known medical history of hospitalization due to COVID-19 within 3 months before screening (V1);
  4. Subjects who had COVID-19 infection before screening (V1) and had not fully recovered to participate in clinical trial operations.
* Suffering from other respiratory diseases simultaneously: α- 1. Antitrypsin deficiency, primary ciliary dyskinesia, lung cancer; Respiratory diseases such as active pulmonary infection, pulmonary tuberculosis, Bronchiectasis, Pulmonary fibrosis, pulmonary Sarcoidosis, pulmonary hypertension, etc. with significant clinical significance assessed by the researchers.
* Chest computed tomography (CT) has found clinically significant abnormalities and believes that the abnormalities are not caused by COPD, and the researchers have determined that they have an impact on the trial results or patient safety. If there is no chest CT report within 3 months before visit 1, a chest CT examination must be performed on visit 1.
* Previously underwent pneumonectomy or lung reduction surgery.
* Previously received lung rehabilitation treatment (those who have been stable for 4 weeks before screening and have remained stable during the trial period can be selected).
* Received oral steroids or roflumilast treatment for COPD within 3 months before screening (Visit 1), or received oral theophylline and/or theophylline derivatives treatment for COPD within 1 months before screening (V1).
* Use non-selective oral administration β Receptor blockers.
* Previously received treatment with ensifentrine and HRS-9821.
* Patients receiving immunotherapy (such as Azathioprine and Cyclophosphamide) within 4 weeks before the screening period.
* The researcher evaluated that during the screening and treatment stages of this study, patients were unable to discontinue the prohibited drugs specified in the protocol.
* The patient has a history of diseases that cannot be controlled at present, including but not limited to diseases of endocrine, thyroid, nervous system, liver, gastrointestinal tract, kidney, blood, Urinary system, immunology or ophthalmic diseases which the investigator judges are clinically significant.
* History or current evidence of cardiovascular diseases with clinical significance. It is defined as any disease that the investigator believes will endanger the safety of patients when participating in the study, or any disease that may affect the effectiveness or safety analysis if the disease/condition worsens during the study; Subjects who have experienced any of the following conditions during visit 1 will be excluded:

  1. myocardial infarction, unstable angina, or stroke within the past 6 months;
  2. There have been unstable or life-threatening arrhythmia requiring intervention within the past 3 months;
  3. New York Heart Association (NYHA) III-IV Heart Failure.
* Have unstable or uncontrollable hypertension.
* Major surgery (requiring general anesthesia) was performed within 8 weeks before the screening visit (V1), or the patient did not fully recover from the surgery during the screening visit (V1), or surgery was planned before the end of the study.
* A history of cured or uncured malignant tumors in any organ or system in the past 5 years.
* Intolerance or allergy to Salbutamol or TQC3721.
* Those who require oxygen therapy, even occasionally.
* Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study.
* Persons who have received live attenuated vaccine within 28 days before randomization, Inactivated vaccine within 7 days, or who plan to receive vaccination during the study period.
* Have a history of drug or alcohol abuse within the past 3 years.
* Individuals who have participated in any clinical trial of drugs or medical devices within 4 weeks or 5 drug half-lives (whichever is longer) prior to screening.
* The researcher believes that there are other situations that are not suitable for participation in the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
The peak of Forced Expiratory Volume in the 1st second (FEV1) (4 weeks) | From baseline to four weeks after treatment.
  Change of the maximum value of FEV1 from baseline to four weeks after treatment

SECONDARY OUTCOMES:
Morning trough FEV1 | From baseline to four weeks after treatment.
  The FEV1 before administration
Average FEV1 (4 weeks) | From baseline to four weeks after treatment.
  Average FEV1 of 3 hours, 12 hours, 24 hours, 0-12 hours and 12-24 hours after administration.
Changes in FEV1 | From baseline to four weeks after treatment.
  Changes in FEV1 at each time point within 24 hours after administration
COPD Assessment Test (CAT) | From baseline to four weeks after treatment.
  Change From Baseline to four weeks after treatment. The score range is 0 to 40 points (0 to 10 is minor influence; 11 to 20 are moderate; 21 to 30 are classified as severe impact; 31 to 40 is very severe).
Modified Medical Research Council (mMRC) Dyspnea Scale Score | From baseline to four weeks after treatment.
  Change From Baseline to four weeks after treatment in mMRC Scoring. The questionnaire is mainly used to evaluate the degree of respiratory distress in patients with chronic obstructive pulmonary disease. According to the symptoms of respiratory distress, the questionnaire is divided into 5 levels, with 0-1 points as less symptoms and ≥ 2 points as more symptoms.
The peak of FEV1 (two weeks) | From baseline to two weeks after treatment.
  Change of the maximum value of FEV1 from baseline to two weeks after treatment
Trough FEV1 | From baseline to two weeks after treatment.
  Change of trough FEV1 from baseline to two weeks after treatment.
Average FEV1 within 3 hours | From baseline to two weeks after treatment
  Average FEV1 within 3 hours after administration
Frequency of Rescue medication | From baseline to four weeks after administration.
  Frequency of Rescue medication used group during the study in the experimental compared to that in the placebo group.
Plasma drug peak concentration (Cmax) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  Plasma drug peak concentration after administration.
Time to maximum concentration (Tmax) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  Time to maximum concentration (Tmax) after administration.
Area Under Curve (AUC) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  Area under the drug concentration-time curve.
Elimination half-life (t1/2) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  Apparent terminal elimination half-life after drug administration.
Apparent volume of distribution (Vd) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  Apparent volume of distribution after drug administration.
Clearance (CL) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  The total drug clearance rate of liver, kidney, etc.
Plasma concentration at steady state (Cav, SS) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  The plasma concentration at which the rate of administration and rate of elimination are in equilibrium.
Minimum concentration (Cmin) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  Plasma drug minimum concentration after administration.
Degree of fluctuation (DF) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  The ratio of the difference between Cmax,ss and Cmin,ss to Cav,ss.
Steady state volume of distribution (Vss) | Within 60 minutes before administration on Day 1, to 24 hours after administration on Day 28.
  Steady state volume of distribution after administration.
Number of cases of adverse events | From baseline to four weeks after treatment.
  Number of cases of adverse events assessed by Common Terminology Criteria for Adverse Events ( CTCAE ) v5.0.
Incidence of adverse events | From baseline to four weeks after treatment.
  Incidence of adverse events assessed by Common Terminology Criteria for Adverse Events ( CTCAE ) v5.0.
Number of cases of serious adverse events. | From baseline to four weeks after treatment.
  Number of cases of serious adverse events assessed by Common Terminology Criteria for Adverse Events ( CTCAE ) v5.0.
Incidence of serious adverse events. | From baseline to four weeks after treatment.
  Incidence of serious adverse events assessed by Common Terminology Criteria for Adverse Events ( CTCAE ) v5.0.
Number of cases of adverse events related to study drug. | From baseline to four weeks after treatment.
  Number of cases of adverse events related to study drug assessed by CTCAE v5.0.
Incidence of adverse events related to study drug. | From baseline to four weeks after treatment.
  Incidence of adverse events related to study drug assessed by CTCAE v5.0.
The peak of FEV1 (Day 1). | From baseline to Day 1.
  Change of the maximum value of FEV1 from baseline to Day 1.
The peak of FEV1 (Day 1 to 4 weeks) | From Day 1 to four weeks after treatment.
  Change of the maximum value of FEV1 from Day 1 to four weeks after treatment
Average FEV1 (Day 2) | From baseline to 24 hours after first treatment.
  Average FEV1 of 3 hours, 12 hours, 24 hours, 0-12 hours and 12-24 hours after administration.
Average FEV1 (Day 1 to 4 weeks) | From Day 1 to four weeks after treatment.
  Average FEV1 of 3 hours, 12 hours, 24 hours, 0-12 hours and 12-24 hours after administration.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Wuhan Sixth Hospital, Wuhan, Hubei
  - Changsha Third Hospital, Changsha, Hunan
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - People's Hospital of Jiangxi province, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang